CLINICAL TRIAL: NCT07170514
Title: Electrical Impedance Tomography vs Dynamic Compliance Guided Positive End-expiratory Pressure Titration During Laparoscopic Gynecological Surgery: A Multi-center, Prospective Randomized Trial - TITRANT
Brief Title: EIT vs Dynamic Compliance Guided PEEP Titration During Laparoscopic Gynecological Surgery
Acronym: TITRANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pest County Flór Ferenc Hospital (Other)
Collaborators: Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged (Other Government); Semmelweis University (Other)
Responsible Party: Principal Investigator, Zoltan Ruszkai, MD, PhD, Head of Department of Anesthesiology and Intensive Therapy, Pest County Flór Ferenc Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BM/8893-3/2025
Record Dates: First submitted 2025-08-29; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Power; Postoperative Pulmonary Complications (PPCs); Oxygenation
Keywords: electrical impedance tomography; dynamic pulmonary compliance; positive end-expiratory pressure; mechanical power; pulmonary protective ventilation; Pao/FiO2; postoperative pulmonary complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-GROUP (Experimental): EIT-guided PEEP titration procedure to achieve individually optimal level of PEEP
  Interventions: Procedure: EIT-guided PEEP titration
- Cdyn-GROUP (Active Comparator): Cdyn-guided PEEP titration procedure to achieve individually optimal level of PEEP
  Interventions: Procedure: Cdyn-guided PEEP titration

INTERVENTIONS:
Procedure: EIT-guided PEEP titration — During the PEEP titration procedure, PEEP will be decreased from 18 cmH2O by 2 cmH2O every 20 ventilatory cycles, until a final PEEP of 6 cmH2O.
  On each level of PEEP EIT parameters and Cdyn values will be recorded in both groups.
  In the EIT-GROUP optimal PEEP is considered as the intersect between the lower percentage of overdistension and collapse, based on the diagnostic tool of the EIT device.
  Arms: EIT-GROUP
Procedure: Cdyn-guided PEEP titration — During the PEEP titration procedure, PEEP will be decreased from 18 cmH2O by 2 cmH2O every 20 ventilatory cycles, until a final PEEP of 6 cmH2O. On each level of PEEP EIT parameters and Cdyn values will be recorded in both groups.
  In the Cdyn-GROUP optimal PEEP is considered as the PEEP value resulting the highest possible Cdyn measured by the ventilator.
  Arms: Cdyn-GROUP

SUMMARY:
The goal of this randomized controlled clinical trial is to compare the pulmonary protective effects of two different positive end-expiratory pressure (PEEP) titrating methods in patients with non-injured lungs undergoing laparoscopic gynecological surgery.

Despite dynamic pulmonary compliance (Cdyn) guided lung protective ventilation has several proven advantages, the investigators hypothesize that optimizing intraoperative mechanical ventilation using electrical impedance tomography (EIT) may further improve patient outcomes, enhance postoperative recovery, shorten in-hospital stay and reduce healthcare related costs.

The main questions aim to answer are:

* May EIT-guided PEEP titration reduce the mechanical power of ventilation and improve oxygenation more significantly than the Cdyn-guided method?
* What effect might a decrease in mechanical power of ventilation have on postoperative pulmonary complications?

Participants will:

* Receive an EIT-guided or a Cdyn-guided PEEP titration procedure during laparoscopic gynecological surgery.
* Be assessed for mechanical power of ventilation, oxygenation, atelectasis and postoperative pulmonary complications during and 2 days after surgery.
* Be followed-up for mortality until the 28th postoperative day.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of two different - electrical impedance tomography guided (EIT) versus dynamic pulmonary compliance guided (Cdyn) - positive end-expiratory pressure (PEEP) titrating methods on mechanical power of ventilation (MP), oxygenation, respiratory mechanics parameters, global inhomogeneity index (GI), overdistension/collapse (ODCL) and postoperative pulmonary complications (PPCs) in patients with non-injured lungs undergoing laparoscopic gynecological surgery. Despite Cdyn-directed lung protective ventilation has several proven advantages, the investigators hypothesize that optimizing intraoperative mechanical ventilation using EIT may further improve patient outcomes by reducing MP responsible for ventilator induced lung injury (VILI) and consequent PPCs. These anticipated advantages may improve the knowledge about individualized intraoperative protective ventilation, enhance postoperative recovery, shorten in-hospital stay and reduce healthcare related costs.

A total number of 200 patients scheduled for laparoscopic gynecological surgery will be enrolled in this study. An equal number of patients will be randomized into the PEEP-EIT and PEEP-Cdyn groups.

Patients randomized into the PEEP-EIT group receive a decremental PEEP titration procedure directed by EIT PEEP Trial of the Dräger PulmoVista 500 device in order to determine the individually optimal level of PEEP (PEEPopt). Patients in the PEEP-Cdyn Group will undergo the same decremental PEEP titration procedure directed by Cdyn measured by the ventilator of the anesthesia workstation.

During the PEEP titration procedure PEEP will be decreased from 18 cmH2O by 2 cmH2O every 20 ventilatory cycles, until a final PEEP of 6 cmH2O. On each level of PEEP Cdyn values will be recorded. In the PEEP-EIT Group PEEPopt is considered as the intersect between the lower percentage of overdistension and collapse, based on the diagnostic tool of the EIT device. In the PEEP-Cdyn Group optimal PEEP is considered as the PEEP value resulting the highest possible Cdyn measured by the ventilator After the titration procedure, a lung protective mechanical ventilation (LPV) will be performed using PEEPopt and low tidal volumes (TV=6 mL/kg, Ideal Body Weight) in both groups.

Mechanical Power, driving pressure, Cdyn, tidal volume in region of interest 3 and 4 (TVROI3, TVROI4) and end-expiratory lung volumes will be recorded immediately after the PEEP titration trial and every 15 minutes during surgery in both groups.

Oxygenation and dead space fraction indicated by the ratio of arterial oxygen partial pressure to fraction of inspired oxygen (PaO2/FiO2) and arterial to end-tidal carbon dioxide difference, respectively, will be recorded every 30 minutes during surgery in both groups. PaO2/FiO2 ratio will be recorded immediately after extubation and 30 mins, 2, 6, 12, 24 and 48 hours after surgery also.

GI and ODCL will be evaluated retrospectively after surgery using the EIT Diag SW 1.6 diagnostic software for Dräger PulmoVista 500.

During the first and second postoperative days EIT measurements will be performed for atelectasis, while arterial blood gas samples will be assessed to screen gas exchange parameters and laboratory examinations will be performed for Sequential Organ Failure Assessment (SOFA) Scores indicating patients' postoperative clinical conditions.

A follow-up period will be performed for mortality until the 28th day after surgery.

ELIGIBILITY:
Inclusion criteria:

* Patient scheduled for elective laparoscopic gynaecological surgery
* Age > 18 years
* Signed consent to participate in the trial

Exclusion criteria:

* Age < 18 years
* American Society of Anesthesiologists (ASA) physical status IV
* History of severe restrictive or chronic obstructive pulmonary disease (COPD, Global Initiative for Chronic Obstructive Lung Disease grades III or IV)
* Uncontrolled bronchial asthma
* Pulmonary metastases
* History of any thoracic surgery
* Need for thoracic drainage before surgery
* Congestive heart failure (NYHA grades III or IV)
* Extreme obesity (BMI>35 kg m-2)
* Lack of patient's consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power (MP) | During surgery
  MP is calculated using a comprehensive formula for volume-controlled ventilator mode:
  MP = 0.098 x RR x TV (L) x [ Ppeak - ½ x (Pplat - PEEP)]
  (RR: respiratory rate TV: tidal volume Ppeak: airway peak pressure Pplat: plateau pressure PEEP: positive end-expiratory pressure)

SECONDARY OUTCOMES:
Oxygenation | From the beginning of surgery to 48 hours after surgery
  Oxygenation indicated by the PaO2/FiO2 ratio
Positive end-expiratory pressure (PEEP) | During surgery
  The level of individually optimal PEEP determined during a PEEP titration procedure
Dynamic pulmonary compliance (Cdyn) | During surgery
  Dynamic pulmonary compliance measured by the ventilator during mechanical ventilation
Driving pressure (dP) | During surgery
  Driving pressure - as an important safety limit of mechanical ventilation - is calculated using a formula:
  dP = Pplat - PEEP
  (Pplat: plateau pressure, PEEP: positive end-expiratory pressure)
Postoperative Pulmonary Complications (PPCs) | From the end of surgery to 48 hours
  PPCs are defined as:
  1. atelectasis detected on computed tomography or chest radiograph,
  2. pneumonia,
  3. Acute Respiratory Distress Syndrome,
  4. pulmonary aspiration (clear clinical history AND radiological evidence) within 48 hours after surgery

OTHER OUTCOMES:
Length of hospital stay | From the date of surgery until discharge, up to 28 days
  Length of hospital stay in days after surgery
In-hospital mortality | From date of surgery until the date of death, up to 28 days
  Death occured during hospital stay after surgery
28-days mortality | 28 days after surgery
  Death occured during 28 days after surgery
Adverse events related to the PEEP titrating procedure | During surgery
  Adverse Events (AEs) related to the PEEP titrating procedure are defined as: severe or prolonged hypotension (systolic blood pressure < 90 mmHg); significant cardiac arrhythmias
  Serious adverse events (SAEs) related to the PEEP titrating procedure are defined as: severe barotrauma leading to pneumothorax; significant prolongation of hospitalization; persistent or significant disability or incapacity; severe deterioration (life-threatening state or even death)

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Ruszkai, MD, PhD, Study Director — Flór Ferenc Hospital Kistarcsa
Locations (3):
- Hungary (3):
  - Semmelweis Hospital Kiskunhalas, Kiskunhalas, Bács-Kiskun county
  - Flór Ferenc Hospital Kistarcsa, Kistarcsa, Pest County
  - Semmelweis University, Budapest

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT07170514/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT07170514/ICF_001.pdf